CLINICAL TRIAL: NCT06681194
Title: A Comparative Study of Silver Nitrate, Triamcinolone, and Their Successive Combined Use on Hypergranulation Tissue in Traumatic Wounds: A Randomized Control Trial
Brief Title: Silver Nitrate vs. Triamcinolone for Treatment of Hypergranulation Tissue
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Francesco Egro (Other)
Responsible Party: Sponsor-Investigator, Francesco Egro, Associate Professor, Plastic Surgery, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY24070165
Record Dates: First submitted 2024-11-06; First posted 2024-11-08 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-11

CONDITIONS: Wound Healing; Granulation Tissue
MeSH Terms: interventions — Silver Nitrate; Triamcinolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Triamcinolone only (Active Comparator): Patients in the triamcinolone group receive triamcinolone 0.5% applied topically to the hypergranulation tissue during their inpatient stay. Upon discharge, patients continue with the same triamcinolone 0.5% treatment, applying it once daily to affected areas in the outpatient setting. Treatment continues until either resolution of hypergranulation tissue (typically within 3-4 weeks) or until 8 weeks have passed without resolution, at which point the patient is considered a treatment failure if open areas persist. Standard wound care practices including appropriate dressings and antibiotics are maintained throughout the treatment period.
  Interventions: Drug: triamcinolone
- Silver nitrate only (Active Comparator): During the inpatient phase, patients in this group receive treatment with silver nitrate sticks applied directly to the hypergranulation tissue. Upon discharge, patients transition to using 0.5% silver nitrate solution for outpatient care, which is applied once daily to the affected areas. The switch to solution form for outpatient treatment is made because it is less painful and easier to apply, particularly on difficult-to-access areas of the body. Treatment continues until either resolution of hypergranulation tissue (typically occurring within 3-4 weeks) or until 8 weeks have passed without resolution, at which point the patient is considered a treatment failure if open areas persist. Throughout the treatment period, standard wound care practices including appropriate dressings and antibiotics are maintained.
  Interventions: Drug: Silver Nitrate
- Combination group (Experimental): The combination group receives treatment with silver nitrate sticks applied directly to the hypergranulation tissue during their inpatient stay. Upon discharge, patients switch from silver nitrate to triamcinolone 0.5%, which they apply once daily to affected areas in the outpatient setting. This treatment continues until either resolution of hypergranulation tissue (typically within 3-4 weeks) or until 8 weeks have passed without resolution, at which point the patient is considered a treatment failure if open areas persist. Standard wound care practices including appropriate dressings and antibiotics are maintained throughout. This combination approach aims to leverage both the initial cauterizing and antimicrobial effects of silver nitrate with the subsequent anti-inflammatory benefits of triamcinolone.
  Interventions: Drug: Silver nitrate + triamcinolone

INTERVENTIONS:
Drug: Silver Nitrate — See "Silver nitrate only" study arm
  Arms: Silver nitrate only
Drug: triamcinolone — See "Triamcinolone only" study arm
  Arms: Triamcinolone only
Drug: Silver nitrate + triamcinolone — See "Combination group" study arm
  Arms: Combination group

SUMMARY:
This randomized controlled trial aims to compare the efficacy of silver nitrate, triamcinolone, and a successive use of both treatments in managing hypergranulation tissue in traumatic wounds. Conducted over a four-year period at UPMC Mercy, the study will involve patients presenting with hypergranulation tissue. Participants will be randomly assigned to receive either topical silver nitrate, topical triamcinolone, or a combination of the two in succession. The study will assess treatment outcomes based on the reduction or resolution of hypergranulation tissue, with the goal of identifying the most effective therapeutic approach. This research will provide valuable insights into optimizing treatment strategies for hypergranulation tissue in traumatic wounds.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years or older.
* Patients must be admitted to the institution with non-infected, traumatic wounds exhibiting hypergranulation tissue.
* Patients must provide consent to participate in the study.
* Eligible wounds include superficial or partial-thickness wounds.
* Wounds will be categorized based on size and depth, with variations controlled for in the statistical analysis.

Exclusion Criteria:

* Patients with known allergies or contraindications to silver nitrate or triamcinolone.
* Patients with wounds that do not exhibit hypergranulation tissue.
* Patients with wounds not primarily due to traumatic injury (e.g., surgical wounds, pressure ulcers).
* Full-thickness, infected, or complex wounds will be excluded, as these may require different management strategies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction in Hypergranulation Tissue Size | From enrollment to 1 year after resolution of hypergranulation
  The investigators will report the changes in hypergranulation tissue size, assessing the change from baseline to follow-up. This will include measuring the hypergranulation size and tracking the percentage reduction over time for participants, with photographic documentation taken at baseline, resolution, and up to one year post-resolution to visually compare size changes. The outcome will evaluate the efficacy of each treatment through clinical observation and standardized wound assessment tools, ensuring that volume is documented as a distinct entry to comply with reporting requirements.
Vancouver Scar Scale (VSS) | From enrollment to 1 year after resolution of hypergranulation
  The scale measures scar characteristics based on color, pliability, height, and area. The VSS consists of three components: 1) Color (0-3), 2) Pliability (0-3), and 3) Height (0-3), with a total area score calculated based on the size of the scar. The overall score ranges from 0 to 13, where 0 indicates normal skin and higher scores represent worse scar quality. Specifically, higher values in color, pliability, and height indicate more severe scarring, while the area score provides an additional measure of size. The individual scores for color, pliability, and height can be summed to compute the total score, with the area score added to provide a comprehensive assessment of scar severity.
Time to healing | From enrollment to 1 year after resolution of hypergranulation
  This outcome records the duration required for the wound to reach significant improvement or closure, helping to assess the treatment's efficiency.
Patient and Observer Scar Assessment Scale (POSAS) | From enrollment to 1 year after resolution of hypergranulation
  The scale measures the quality of scars from both patient and observer perspectives. The scale includes two main components: the Patient Scale and the Observer Scale. Each component consists of 6 items rated on a scale from 1 to 10, where 1 represents "no scar" and 10 represents "the worst scar imaginable," allowing for a total score range of 6 to 60 for each scale. Higher scores indicate worse outcomes, reflecting greater scar severity and patient distress. To compute a total score, the subscale scores can be summed, providing an overall assessment of scar quality from both perspectives.

SECONDARY OUTCOMES:
Cutometry | From enrollment to 1 year after resolution of hypergranulation
  This outcome assesses the structural integrity of the skin post-treatment, measured using a cutometer. The cutometer evaluates skin firmness and elasticity by applying a vacuum to the skin and measuring the degree of deformation. This assessment provides quantitative data on how well the skin maintains its structure after hypergranulation treatment, allowing for a comparison of improvements over time.
Scar color | From enrollment to 1 year after resolution of hypergranulation
  Using colorimetry, this outcome measures changes in skin/scar color, providing insights into the effects of the treatments on skin appearance.
Treatment satisfaction | From enrollment to 1 year after resolution of hypergranulation
  The satisfaction scale for evaluating hypergranulation treatment uses a numeric scale from 1 to 10, where respondents indicate their level of satisfaction with the treatment. A score of 1 represents "Very Dissatisfied," indicating complete unhappiness with the treatment, while a score of 10 signifies "Completely Satisfied," reflecting total contentment with the treatment and its outcomes. This scale allows patients to provide a clear, quantifiable assessment of their treatment experience, which can inform improvements in care and patient outcomes.
Complications | From enrollment to 1 year after resolution of hypergranulation
  This outcome will report the number of participants experiencing any complications related to hypergranulation treatment, including infection, skin sloughing, and delayed wound healing. By tracking these complications, the investigators will evaluate the safety profile of each treatment method. Specifically, the investigators will document the incidence of each complication, providing a clear metric for assessing the overall safety and tolerability of the treatments used. This information will be crucial for understanding the risks associated with each approach and guiding future treatment decisions.
Numeric Rating Scale (NRS) | From enrollment to 1 year after resolution of hypergranulation
  The Numeric Rating Scale (NRS) for pain is a subjective measure used to assess a patient's level of pain on a scale from 0 to 10. Patients are asked to rate their pain by selecting a number that best represents their current pain level. This scale allows healthcare providers to quickly gauge the severity of pain and monitor changes over time, facilitating appropriate pain management strategies.
Durometry | From enrollment to 1 year after resolution of hypergranulation
  The mechanical properties of the skin will be evaluated using a durometer, which measures the hardness of the skin. This measurement reflects the skin's resilience and texture following treatment. By documenting changes in skin hardness, the investigators can gain insights into how the treatment affects the skin's overall quality and tactile properties, contributing to a comprehensive understanding of treatment efficacy.
Elastometry | From enrollment to 1 year after resolution of hypergranulation
  Skin elasticity will be assessed using an elastometer, which quantifies the skin's ability to stretch and return to its original shape. This outcome reflects improvements in the skin's mechanical properties and overall health post-treatment. By analyzing the elasticity of the skin, the investigators can better understand the treatment's impact on skin recovery and resilience, providing valuable information for patient care and outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco M Egro, MD, MSc, MRCS, Principal Investigator — Department of Plastic Surgery, University of Pittsburgh Medical Center
Locations (1):
- UPMC Mercy Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
The investigators may provide deidentified patient information journals if requested; however, the investigators are currently undecided about the likelihood of such requests. While the investigators recognize the importance of data sharing for advancing research, the investigators must consider patient confidentiality and ethical considerations when determining the approach.

REFERENCES:
- [Background] Moio M, Mataro I, Accardo G, Canta L, Schonauer F. Treatment of hypergranulation tissue with intralesional injection of corticosteroids: preliminary results. J Plast Reconstr Aesthet Surg. 2014 Jun;67(6):e167-8. doi: 10.1016/j.bjps.2014.03.017. Epub 2014 Mar 26. No abstract available. PMID 24725728
- [Background] Baumann ME, DeBruler DM, Blackstone BN, Coffey RA, Boyce ST, Supp DM, Bailey JK, Powell HM. Direct comparison of reproducibility and reliability in quantitative assessments of burn scar properties. Burns. 2021 Mar;47(2):466-478. doi: 10.1016/j.burns.2020.07.018. Epub 2020 Aug 2. PMID 32839037
- [Background] McShane DB, Bellet JS. Treatment of hypergranulation tissue with high potency topical corticosteroids in children. Pediatr Dermatol. 2012 Sep-Oct;29(5):675-8. doi: 10.1111/j.1525-1470.2012.01724.x. Epub 2012 May 21. PMID 22612258
- [Background] Linneman PK, Litt J. Hypertrophic Granulation Wounds Treated With Silver Nitrate Sticks or With Topical Steroid: Rate of Wound Closure. J Burn Care Res. 2022 Mar 23;43(2):403-407. doi: 10.1093/jbcr/irab196. PMID 34687202
- [Background] Maynell KB, West W 3rd, Marek J, Wright B, Bodnar M, Le NK, Whalen K, Taylor L, Troy J, Smith D Jr, Laun J. Utilization of Topical Polysporin and Triamcinolone for the Treatment of Hypergranulation Tissue. J Burn Care Res. 2024 May 6;45(3):669-674. doi: 10.1093/jbcr/irad205. PMID 38165005